CLINICAL TRIAL: NCT05586477
Title: Does Diphenhydramine Alter Thermoregulatory Responses During Exercise?
Brief Title: Diphenhydramine and Sweating
Acronym: BENEXE2022
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lakehead University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022509; 265937 (Other: Health Canada, Control Number)
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Diphenhydramine Causing Adverse Effects in Therapeutic Use; Hyperthermia; Allergic Rhinitis; Sweating
Keywords: thermoregulation; diphenhydramine; anticholinergic; sweating
MeSH Terms: conditions — Hyperthermia; Rhinitis, Allergic | interventions — Diphenhydramine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Order (Placebo - Diphenhydramine) (Other): On separate days, participants will march on a treadmill for 60 minutes at a fixed rate of oxygen consumption (~1.75 liters of oxygen consumption per minute) in ~28°C and 30% relative humidity
  Interventions: Drug: Placebo; Drug: Diphenhydramine
- Intervention Order (Diphenhydramine -Placebo) (Other): On separate days, participants will march on a treadmill for 60 minutes at a fixed rate of oxygen consumption (~1.75 liters of oxygen consumption per minute) in ~28°C and 30% relative humidity
  Interventions: Drug: Placebo; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Placebo — A placebo pill (i.e., sugar) will be consumed 2 h before intervention.
Drug: Diphenhydramine — Extra strength Benadryl (DIN 02470144) will be consumed 2 h before intervention

SUMMARY:
In 2012, it was estimated that nearly 1 in 4 Canadians suffer from allergic rhinitis. To add, 78% of individuals working in predisposing environments are predicted to develop occupational rhinitis. Currently, the most popular treatment for rhinitis is antihistamine medication such as diphenhydramine, a first-generation antihistamine sold commercially as Benadryl®. Due it its anticholinergic effects, diphenhydramine has been suggested to impair the whole body sweating response during heat stress, potentially leaving consumers at an increased risk of heat-related illness. This randomized control trial approved by Health Canada will investigate whether ingesting extra strength diphenhydramine (50mg) will alter whole-body sweat losses during 60 minutes of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Able to safely perform ~60 minutes of moderate intensity exercise
* No known hypersensitivity to diphenhydramine
* Not on any prescribed medication
* Body-mass index (BMI) less than 30

Exclusion Criteria:

* Outside 18 - 49 years of age
* Diagnosed with any cardiovascular, respiratory, neurological or metabolic disease
* History of any cardiovascular, respiratory, neurological or metabolic disease
* Unable to exercise for 60 minutes at moderate intensity, or have a musculoskeletal injury
* BMI > or = 30

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Whole body sweat loss | Measured during both placebo and diphenhydramine intervention trials trials, separated by no more than 28 days
  Change in body mass from pre- to post-exercise corrected for respiratory and metabolic water losses using a digital platform scale accurate to +/- 2 grams.

SECONDARY OUTCOMES:
Change in rectal temperature | Measured during both placebo and diphenhydramine intervention trials trials, separated by no more than 28 days
  Change in rectal temperature from pre- to post- exercise using a pediatric grade thermistor

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Ravanelli, PhD, Principal Investigator — Lakehead University
Locations (1):
- Lakehead Unviersity, Thunder Bay, Ontario, Canada

REFERENCES:
- [Derived] Newhouse D, Mihalcin E, Lefebvre K, Nucci M, Ravanelli N. Thermal and Cardiovascular Responses during Exertional Heat Stress after Diphenhydramine Use: A Randomized Crossover Trial. Med Sci Sports Exerc. 2024 Dec 1;56(12):2328-2337. doi: 10.1249/MSS.0000000000003527. Epub 2024 Jul 31. PMID 39140777